CLINICAL TRIAL: NCT05367076
Title: Development of a Web-based Exercise Training Program for Brain Repair and Cognitive Recovery for Paediatric Brain Tumour Survivors in the Community: a Feasibility Study
Brief Title: Fitness to Aid the Brain and Cognitive Skills
Acronym: Fit ABCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Donald Mabbott, Senior Scientist and Program Head, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000073462
Record Dates: First submitted 2022-04-22; First posted 2022-05-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Brain Tumor; Cognitive Impairment
Keywords: Exercise; Physical functioning
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FitABCS exercise (Experimental): Web-based community-led, 12-week exercise program
  Interventions: Behavioral: Web-based Aerobic Exercise Program
- FitABCS control (No Intervention): Healthy control

INTERVENTIONS:
Behavioral: Web-based Aerobic Exercise Program — Community based FTTs will use a web-based platform to deliver a 12-week exercise training program (120-minute group sessions of aerobic activity 3 times/week). Each session will include:
  * Warm-up activities
  * Aerobic activities and fitness training in a game-like fashion
  * Organized sports/games
  * Cool down activity
  * Snack/reward time
  Arms: FitABCS exercise

SUMMARY:
The study will assess the feasibility of a pilot clinical trial of community-led aerobic exercise training for paediatric brain tumour survivors (PBTS) and the feasibility of a web-based platform to deliver this exercise training. It is hypothesized that 12 weeks of community-led exercise training will be feasible for PBTS and the web-based platform will be feasible to deliver exercise training by community-based instructors.

DETAILED DESCRIPTION:
PBTS will complete 12 consecutive weeks of exercise training. Exercise training will involve 90-minute group sessions of aerobic activity 3 times/week with a 30-minute snack/reward time. The investigators anticipate participants will complete the exercise training program in cohorts, each comprised of a minimum of 3 and maximum of 10 participants. With a minimum of 3 participants per cohort, in order for us to achieve the investigators' goal of recruiting 30 participants, the investigators anticipate running approximately 7 cohorts. Participants will be assigned to a cohort based on proximity to session location and availability to attend sessions.

Site Description:

This is a single-site trial, as participants will be recruited from SickKids. Community-led exercise training will be delivered at various locations across the Greater Toronto and Hamilton Area (GTHA). Exercise training sessions will be conducted in partnership with Wellspring, a network of community support services across the GTHA for individuals diagnosed and treated for cancer. The investigators have developed a web-based platform for Fitness Trainers/Therapists (FTTs) to i) educate them on working with PBTS, ii) build exercise session plans, and iii) provide feedback on sessions and overall web-based platform functionality and usability. The web-based platform will allow the administration of community-led exercise training in any location. To test the feasibility of the web-based platform, the investigators will be administering exercise training in approximately 5 locations associated with Wellspring centres (and/or surrounding gymnasiums or outdoor space) and Wellspring FTTs.

Study Intervention Description:

Exercise training will consist of group sessions of aerobic exercise. Each session will include five (5) components:

1. Warm-up activities
2. Aerobic training activities
3. Group sports/games
4. Cool-down activities
5. Snack/reward time The goal of the intervention is to increase and maintain participants' heart rate for at least 30 minutes per session at a minimum of 80% of participants' peak heart rate achieved during a baseline fitness assessment. Increased heart rate will mainly take place during the aerobic circuit training and group sport/game components of each session. Heart rate will be measured using heart rate monitors.

Description of study population:

* Sample size: n = 40 (30 PBTS, 10 Healthy Controls)
* Age: 6-17 years
* Sex: males and females
* General health [PBTS]: Patients who have completed treatment for hemispheric or posterior fossa tumours and do not have severe neurological/motor dysfunction that would preclude safe participation in an exercise program
* General health [Healthy Controls]: Do not have neurological/motor dysfunction that would preclude safe participation in baseline assessment or have a prior history of neurodevelopmental or neurological disorder, cerebral palsy, developmental delay or learning disability at time of enrollment
* Geographic location: Canada

ELIGIBILITY:
Inclusion Criteria:

1. Between 6 years and 17 years and 11 months of age at time of enrollment
2. Diagnosed with a brain tumour
3. 1 to 15 years between diagnosis and time of study enrollment
4. Medically stable (i.e. must be in remission) as determined by a permanent SickKids staff Neuro-Oncologist
5. Either declare English as their native language or have at least two years of schooling in English at the time of their first assessment
6. Have a parent or legal guardian willing to complete the Health and Quality of Life measures
7. Informed consent (and assent, where applicable) will be obtained from the participants and/or their legal guardians

Exclusion Criteria:

1. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate, interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk
2. Diagnosed with a neurodevelopmental or neurological disorder, cerebral palsy, developmental delay or learning disability prior to initial brain tumour diagnosis that would preclude safe participation
3. Receiving palliative care
4. Require sedation for neuroimaging
5. Have ferrous metal implants (i.e. cochlear implant, braces, etc.)
6. Have a programmable shunt
7. Pregnant
8. Completed any prior cognitive rehabilitation intervention within three months of enrollment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of the exercise program: The probability that 30 eligible patients will be recruited | 24 Months
  In order to determine the feasibility of a 12 weeks of community-led exercise training for PBTS, there will be satisfactory patient recruitment. The goal is to recruit n=30 participants (≥25% probability)
  Measure: The Bayesian probability statistic that 30 eligible patients will be recruited
Feasibility of the exercise program: The probability that a recruited participant will attend ≥60% of exercise training sessions | 24 weeks
  In order to determine the feasibility of a 12 weeks of community-led exercise training for PBTS, there will be satisfactory participant attendance. The goal is for a participant to attend ≥60% of exercise training sessions (≥80% probability of participants).
  Measure: The Bayesian probability statistic that participants will rate the therapeutic alliance between participant/instructor as cooperative and collaborative.
Feasibility of the exercise program: The probability that a recruited participant will complete all study procedures | 24 weeks
  In order to determine the feasibility of a 12 weeks of community-led exercise training for PBTS, there will be satisfactory participant adherence to study procedures (neuroimaging, cognitive, health and quality of life (QOL), cardiovascular fitness and physical functioning assessments). The goal is for a recruited participant to complete all study procedures (≥80% probability).
  Measure: The Bayesian probability statistic that a recruited participant will complete all study procedures
Feasibility of the exercise program: The probability that instructors will adhere to the web-based platform to deliver exercise training | 24 weeks
  In order to determine the feasibility of a 12 weeks of community-led exercise training for PBTS, there will be satisfactory instructor adherence to deliver the program. The goal is for instructors to adhere to the web-based platform to deliver exercise training (≥80% probability).
  Measure: The Bayesian probability statistic that instructors will adhere to the web-based platform to deliver exercise training
Feasibility of the exercise program: The probability that instructors will develop a therapeutic alliance with the participants | 24 weeks
  In order to determine the feasibility of a 12 weeks of community-led exercise training for PBTS, there will be satisfactory rating by the participant of the therapeutic alliance between participants and instructors. The goal is for participants to have a cooperative and collaborative relationship with the instructors, as rated by the Therapeutic Alliance Scales for Children-Revised questionnaire.
  Measure: The Bayesian probability statistic that the therapeutic alliance between participant/instructor will be comparable across cohorts.
Feasibility of the web-based platform: The probability that instructors will rate the platform as acceptable | 24 weeks
  In order to determine the feasibility of a web-based platform to be used by community-based FTTs to deliver exercise training to PBTS, instructors will rate the platform as acceptable (e.g. would recommend to others, would continue to use). The goal is for instructors to rate the the platform as acceptable, indicating ease of use and satisfaction (≥80% probability).
  Measure: The Bayesian probability statistic that instructors will rate the platform as acceptable
Feasibility of the web-based platform: The probability that instructors will rate the platform as relevant | 24 weeks
  In order to determine the feasibility of a web-based platform to be used by community-based FTTs to deliver exercise training to PBTS, instructors will rate the platform as relevant (e.g. includes all necessary components to administer an exercise program, would choose to use such a tool to deliver an exercise program).The goal is for the instructors to rate the platform as relevant, indicating the presence of necessary information (≥80% probability).
  Measure: The Bayesian probability statistic that instructors will rate the platform as relevant
Feasibility of the web-based platform: The probability that instructors will rate the platform as efficient | 24 weeks
  In order to determine the feasibility of a web-based platform to be used by community-based FTTs to deliver exercise training to PBTS, instructors will rate the platform as efficient (e.g. is useful). The goal is for the instructors to rate the platform as efficient, indicating its usefulness (≥80% probability).
  Measure: The Bayesian probability statistic that instructors will rate the platform as efficient

OTHER OUTCOMES:
Comparison of community-led vs. historical hospital-led exercise training program: Changes in hippocampal volume | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training for PBTS in terms of changes in hippocampal volume using MRI (magnetic resonance imaging).
  Measures: Anatomical T1 weighted MRI will acquire estimates of hippocampal volume
Comparison of community-led vs. historical hospital-led exercise training program: Changes in neural communication | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training for PBTS in terms of changes in neural communication, as estimated by functional connectivity during magnetoencephalography (MEG) recording.
  Measures: The weighted phase lag index (wPLI) will be used to measure functional connectivity during MEG recording as an estimate of neural communication
Comparison of community-led exercise training to historical data from a hospital-led exercise training program: Changes in information processing speed | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training program for PBTS in terms of changes in information processing speed.
  Measure: Scores on the Rapid Visual Information Processing subtest of the Cambridge Neuropsychological Test Automated Battery
Comparison of community-led exercise training to historical data from a hospital-led exercise training program: Changes in controlled attention | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training program for PBTS in terms of changes in controlled attention.
  Measure: Scores on the Match to Sample Visual Search Task subtest of the Cambridge Neuropsychological Test Automated Battery
Comparison of community-led exercise training to historical data from a hospital-led exercise training program: Changes in declarative memory | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training program for PBTS in terms of changes in declarative memory.
  Measures: Scores on the Delayed Matching to Sample Task subtest of the Cambridge Neuropsychological Test Automated Battery
Comparison of community-led exercise training to historical data from a hospital-led exercise training program: Changes in cardiovascular fitness (heart rate, and sub-maximal and maximal work rates) | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training program for PBTS in cardiovascular fitness, including heart rate, sub-maximal and and maximal work rates.
  Measures: 6-Minute Walk Test and electrically braked cycle ergometer to measure heart rate, and sub-maximal and maximal pro-rated work rates
Comparison of community-led exercise training to historical data from a hospital-led exercise training program: Changes in physical functioning (bilateral coordination and balance, and running speed/agility and strength) | Baseline, Week 13, and Week 25
  To compare community-led exercise training to historical data from a hospital-led exercise training program for PBTS in terms of changes in physical functioning, including bilateral coordination and balance (body coordination), and running speed/agility and strength (strength and agility).
  Measure: Bilateral coordination and balance (body coordination), and running speed/agility and strength (strength and agility) using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition. Minimum points scored: 0, maximum points scored: 80; higher scores account for greater motor proficiency (better outcomes)
Impact of this study intervention on PBTS: Changes in white matter microstructure | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in white matter microstructure using diffusion kurtosis imaging (DKI)
  Measures: DKI will acquire kurtosis measures of water diffusion in the brain (mean, axial, radial kurtosis)
Impact of this study intervention on PBTS: Changes in hippocampal volume | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes hippocampal volume using Anatomical T1 MRI
  Measures: Hippocampal volume estimated using Anatomical T1 MRI
Impact of this study intervention on PBTS: Changes in neural communication | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in neural communication as estimated by functional connectivity during MEG recording.
  Measures: The wPLI will be used to measure functional connectivity during MEG recording as an estimate of neural communication
Impact of this study intervention on PBTS: Changes in information processing speed | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in information processing speed.
  Measures: Scores on the Pattern Comparison Processing Speed Test subtest of the National Institutes of Health Toolbox and Reaction Time Task subtest RTI subtest of the Cambridge Neuropsychological Test Automated Battery
Impact of this study intervention on PBTS: Changes in controlled attention | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in controlled attention
  Measures: Scores on the Flanker Inhibitory Control & Attention Task subtest of the National Institutes of Health Toolbox, and the Stop Signal Task, Rapid Visual Information Processing, and Match to Sample Visual Search subtests of the of the Cambridge Neuropsychological Test Automated Battery
Impact of this study intervention on PBTS: Changes in declarative memory | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in declarative memory
  Measures: Scores on the Children's Auditory Verbal and Learning Test-2 or Rey Auditory Verbal Learning Test (for participants who will be 18 years of age at the time of study completion) and Delayed Matching to Sample subtest of the Cambridge Neuropsychological Test Automated Battery
Impact of this study intervention on PBTS: Changes in full scale intelligence | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in full scale intelligence.
  Measures: Scores on the Vocabulary and Matrix Reasoning subtests of the Wechsler Abbreviated Scale of Intelligence-Second Edition
Impact of this study intervention on PBTS: Changes in MEG behavioural measures | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in MEG behavioural measures.
  Measures: Reaction time and accuracy scores on the Simple and Choice Visual-Motor Reaction Time Task, and Multi-Source Interference Task during MEG recording
Impact of this study intervention on PBTS: Health and QOL | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in health and QOL
  Measure: Scores on the Patient-Reported Outcomes Measurement Information System - Global health 7+2, Pediatric Quality of Life Scale generic core scale, physical activity preference questionnaire and Habitual Physical Activity Scale. All health and QOL measures are parent-proxy reports.
Impact of this study intervention on PBTS: Changes in cardiovascular fitness (heart rate, and sub-maximal and maximal work rates) | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training on the following outcomes in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in cardiovascular fitness, including heart rate, sub-maximal and and maximal work rates.
  Measures: 6-Minute Walk Test and electrically braked cycle ergometer to measure heart rate, and sub-maximal and maximal pro-rated work rates
Impact of this study intervention on PBTS: Changes in physical functioning (bilateral coordination and balance, and running speed/agility and strength, and ataxia) | Baseline, Week 13, and Week 25
  To investigate the impact of community-led exercise training in PBTS to provide preliminary data for a subsequent adequately powered randomized controlled trial in terms of changes in physical functioning, including bilateral coordination and balance (body coordination), and running speed/agility and strength (strength and agility), and ataxia.
  Measure: Bilateral coordination and balance (body coordination), and running speed/agility and strength (strength and agility) using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition. Minimum points scored: 0, maximum points scored: 80; higher scores account for greater motor proficiency (better outcomes), strength assessment conducted by a registered Physiotherapist and the Scale for the Assessment and Rating of Ataxia. Minimum points scored: 0, maximum points scored: 40; higher scores indicate increased severity of ataxia (worse outcome)
Impact of this study intervention on PBTS: Changes in physical functioning as reported by parent (PEDI-CAT) | week 25
  To investigate the impact of community-let exercise training in PBTS to improve physical functioning in the participant's daily life, as reported by their parent.
  Measure: Parent report the ease of physical (and cognitive) activities in their child's daily life.
Comparing brain structure outcomes before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in brain structure following exercise training and at 3-month follow up compared to before exercise training.
  Measures: brain structure (MRI) as assessed through white matter microstructure as estimated by kurtosis (mean, axial, and radial).
Comparing brain function outcomes before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in brain function following exercise training and at 3-month follow up compared to before exercise training.
  Measures: Hippocampal volume and functional connectivity (MEG) as estimated by the weighted Phase Lag Index (wPLI)
Comparing cognitive outcomes (information processing speed) before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in cognition following exercise training and at 3-month follow up compared to before exercise training
  Measures: Pattern Comparison Processing Speed Test, Reaction Time (RTI) (reaction time for simple and 5-choice conditions= measured in milliseconds, shorter reaction time is better)
Comparing cognitive outcomes (controlled attention) before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in cognition following exercise training and at 3-month follow up compared to before exercise training
  Measures: Flanker Inhibitory Control & attention Task, SST, RVP, and MTS)
  SST: Stop Signal Task (stop signal reaction time = milliseconds, lower is better)
  RVP: Rapid Visual information Processing (A prime = range 0-1, higher is better)
  MTS: Match To Sample visual search (correct trials (all trials) = %, higher is better)
Comparing cognitive outcomes (declarative memory) before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in cognition following exercise training and at 3-month follow up compared to before exercise training
  Measures: CAVLT-2 or RAVLT, DMS
  CAVLT-2: Children's Auditory Verbal Learning Test 2 (standard scores range from <60 to >140, higher is better)
  RAVLT: Rey Auditory Verbal Learning Test (T scores range from < 20 to >80, higher is better)
  DMS: Delayed Matching to Sample (correct trials (all trials) = %, higher is better)
Comparing cognitive outcomes (full scale intelligence quotient) before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in cognition following exercise training and at 3-month follow up compared to before exercise training
  Measures: 2 subtests (Vocabulary, Matrix Reasoning) where T-scores are computed (20-80 range) with a higher value denoting a better score.
Comparing cognitive outcomes (MEG behavioral measures) before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in cognition following exercise training and at 3-month follow up compared to before exercise training
  Measures: Go/No-Go task, MSIT
  MSIT: Multi Source Interference Task (reaction time= milliseconds, lower is better; accuracy = /1, higher is better; this also applies to Go/No-Go)
Comparing health outcomes before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in health and quality of life following exercise training and at 3-month follow- up compared to before exercise training.
  Measure: PROMIS parent proxy scale- Global health 7+2, PedsQL generic core parent-proxy report
  PROMIS: Patient-Reported Outcomes Measurement Information System (T-scores range 14.7-68.78, higher is better)
  PedsQL: Pediatric Quality of Life scale (range 0-100, higher score is better QoL)
Comparing quality of life outcomes before and after community-based exercise training to a group of healthy age-matched peers | Baseline
  To investigate whether PBTS participants more closely resemble their healthy peers in health and quality of life following exercise training and at 3-month follow- up compared to before exercise training.
  Measure: HAES parent-proxy report, and PEDI-CAT
  HAES: Habitual Activity Estimation Scale (active hours = higher is better, inactive hours= lower is better)
  PEDI-CAT: pediatric evaluation of disability inventory computer adaptive test (scaled scores range 20-80, higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Donald J Mabbott, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No